CLINICAL TRIAL: NCT00838331
Title: Adverse Effects of RBC Transfusions: A Unifying Hypothesis
Acronym: INOBA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, John D Roback, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00015316
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Volunteers
Keywords: Blood Transfusions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fresh blood, then aged blood (Experimental)
  Interventions: Biological: Fresh blood; Biological: Aged blood

INTERVENTIONS:
Biological: Fresh blood — For fresh transfusions, a whole blood unit will be drawn from volunteers, processed, and then reinfused on the same day during the study. For impaired and repaired transfusions, the volunteers will be brought to the blood bank to donate; then, after processing and the appropriate length of storage (eg, 28 days), they will return for the FBF studies. Since recipients of fresh transfusions are relatively anemic after donation and before reinfusion, recipients of impaired/repaired transfusions should also be mildly anemic for the study. Thus, they will donate another whole blood unit prior to beginning the study course, they will be transfused with their stored unit during the study, and then the autologous unit collected at the beginning of the day will be reinfused at the end of the day after the study is complete.
Biological: Aged blood — In a separate aim, the FMD assay will be used to investigate NO-mediated vasodilation in patients with CVD who are receiving transfusions. Over 60% of blood orders for cardiology patients at Emory are for 2 units or more. Therefore, when a 2-unit order is placed on a consented patient, they will be issued both fresh (< 7 days) and impaired (> 28 days) compatible units from inventory. Prior to starting transfusions, the patient will be randomized to either receive the fresh or the older unit first. All RBC units will be ACD/AS1. Units will also be leukoreduced and/or irradiated, if either of those modifications were found to impair NO bioavailability in prior studies. If washing or rejuvenation were found to be successful in significantly "repairing" NO bioavailability in previous aims, some patients may also receive impaired and repaired (> 28 days; washed or rejuvenated) RBC transfusions.

SUMMARY:
Transfusion of red blood cells is often used in critically ill patients with low red blood cell counts to prevent disease progression and death. Recent studies suggest that the use of "aged" versus "fresh" red blood cells are associated with worse clinical outcomes. There is evidence that red blood cells work with the cells lining our blood vessels to produce a variety of substances that normally cause arteries to relax and increase blood supply. Two of these substances are called nitric oxide (NO) and endothelium-derived hyperpolarizing factor (EDHF). The investigators are trying to determine the nature of these substances in human beings when they are transfused "aged" versus "fresh" red blood cells. It is their thought that "aged" red blood cells have less of the substances (NO and EDHF) that naturally relax our arteries and further changes the blood supply. One way to determine this is to transfuse a subject's own "aged" and "fresh" red blood cells and inject substances such as L-NMMA (L-NG monomethyl arginine) and TEA (tetraethylammonium chloride), which block the production of NO and EDHF respectively, and then, study what happens to the blood flow.

There is evidence that red blood cells produce NO, which normally causes arteries to relax and increase blood supply. The investigators will try to determine the nature of NO in red blood cells and whether the amount of this substance is altered because of different blood processing and storage techniques. It is their thought that "aged" red blood cells have less NO that naturally relaxes our arteries and further changes the blood supply. This study is designed to determine the most ideal way of storing and processing blood.

DETAILED DESCRIPTION:
Transfusion of red blood cells (RBCs) is often effective at preventing morbidity and mortality in anemic patients. In contrast, recent studies indicate that some RBC components may have functional defects ("RBC storage lesions") that actually cause morbidity and mortality when transfused. For example, patients transfused with RBCs stored >14 days have statistically worse outcomes than those receiving "fresher" RBC units. In addition to the age of stored RBCs, the volume transfused may be important. The TRICC study showed that specific patients whose transfusions were limited by a restrictive trigger (RBCs transfusions only when hemoglobin [Hb] < 7 g/dL) had significantly better outcomes than those transfused with a more liberal trigger ([Hb] < 10 g/dL Hb). This finding has been particularly difficult to understand since conventional wisdom suggests that an elevated [Hb] should be beneficial because it supports increased O2 delivery. Recipient-specific factors may also contribute to the occurrence of these adverse events. Unfortunately, these events have been difficult to investigate because up to now they have existed only as "statistical occurrences" of increased morbidity and mortality in large data sets. There are currently no clinical or laboratory methods to detect or study them in individual patients.

The microcirculation is composed of a continuum of small vessels including small arterioles, capillaries, and post-capillary venules. The microcirculation represents an actively-adjusting vascular circuit that matches blood flow (and O2 delivery) to local tissue oxygen demands. While the physiologic mechanisms that match O2 delivery to local requirements are incompletely understood, endothelium-derived nitric oxide (NO) clearly plays an important role. Interestingly, recent work has revealed that in addition to transporting O2 and CO2, the RBC also controls local NO concentrations and thus may also play a surprisingly important role in regulating blood flow in the microcirculation.

Herein, the investigators bring together previously unconnected data to propose a unifying hypothesis, centered on insufficient NO bioavailability (INOBA), to explain the increased morbidity and mortality observed in some patients following RBC transfusion. In this model, variables associated with RBC units (storage time; 2,3-DPG concentration) and transfusion recipients (endothelial dysfunction; hematocrit [Hct]) collectively lead to changes in NO levels in vascular beds. Under certain circumstances, these variables are "aligned" such that NO concentrations are markedly reduced, leading to vasoconstriction, decreased local blood flow and insufficient O2 delivery to end organs. Under these circumstances, the likelihood of morbidity and mortality escalates. The INOBA hypothesis is attractive because of its explanatory power and because it leads to a number of readily testable predictions, which will be investigated in the following aims:

Aim 1: To investigate the effects of blood processing and storage (using standard FDA-approved conditions) on NO production and scavenging by human RBCs/Hb in vitro. Using sensitive biochemical assays (electron spin resonance [ESR]) and a rat aortic ring in vitro bioassay, the investigators will test the effects of RBC storage time, leukoreduction, and irradiation on NO synthesis and/or scavenging by intact RBCs and free Hb. Modifications such as washing and rejuvenation will be investigated as possible approaches to correct abnormalities in NO bioavailability.

Aim 2: To transfuse healthy volunteers and investigate the effects of storage-related RBC changes on blood flow, tissue oxygenation, and biomarkers of cardiovascular function. The investigators will determine whether RBCs prepared and stored under conditions that alter NO bioavailability in vitro (Aim 1) inhibit NO-mediated vasodilation, reduce tissue perfusion, and decrease tissue O2 delivery in healthy transfusion recipients in vivo. The role of 2,3-DPG depletion as well as exercise-induced O2 demand will also be investigated with these specialized experimental systems.

ELIGIBILITY:
Aim 1:

Inclusion Criteria:

* Healthy male or female volunteers (age 21-60 years)

Must meet guidelines for blood donors including:

* standard blood donor history questionnaire
* body weight of at least 110 lbs
* hemoglobin concentration of at least 12.5 gm/dL
* body temperature of no more than 99.5 oF
* pulse of 50-100 bpm
* blood pressure < 180/100
* test negative for the standard battery of blood donor screening tests (anti-HIV, HIV RNA, anti-HCV, HCV RNA, HBsAg, anti-HBc, anti-HTLV-I/II, and WNV RNA)

Aim 1:

Exclusion Criteria:

* Failure to pass the blood donor history questionnaire
* Positive results on the standard battery of blood donor screening tests
* Failure to meet criteria for donation

Aim 2:

Inclusion Criteria:

* Healthy male or female volunteers (age 21-80 years)

Exclusion Criteria:

* Presence of intercurrent illness or other chronic diseases
* Renal failure (creatinine>1.4 mg/dl)
* Pregnancy
* Allergies to aspirin
* Bleeding disorders
* Uncontrolled hypertension with BP > 180 mmHg systolic and > 120 mmHg diastolic
* Acute infection in previous 4 weeks
* History of substance abuse
* Liver failure (Liver enzymes >2x normal)
* Inability to give informed consent
* Inability to return to Emory for follow-up

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-04; Primary Completion 2013-05 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arshed A Quyyumi, MD, Principal Investigator — Emory University; John Roback, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Hayek SS, Neuman R, Ashraf K, Sher S, Newman JL, Karatela S, Roback JD, Quyyumi AA. Effect of storage-aged red blood cell transfusions on endothelial function in healthy subjects. Transfusion. 2015 Nov;55(11):2768-70. doi: 10.1111/trf.13276. No abstract available. PMID 26559401
- [Derived] Neuman R, Hayek S, Rahman A, Poole JC, Menon V, Sher S, Newman JL, Karatela S, Polhemus D, Lefer DJ, De Staercke C, Hooper C, Quyyumi AA, Roback JD. Effects of storage-aged red blood cell transfusions on endothelial function in hospitalized patients. Transfusion. 2015 Apr;55(4):782-90. doi: 10.1111/trf.12919. Epub 2014 Nov 13. PMID 25393772

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Seven subjects withdrew prior to transfusion.
Groups:
- Fresh Blood, Then Aged Blood: Subjects donated one unit of blood, which was processed, stored for 3-5 days, then infused back to the subject (Fresh Blood). At least 8 weeks later, they returned, donated another unit of blood, which was stored for 40-42 days, then infused back to the subject (Aged Blood). Before and after each transfusion, the subjects was tested with a variety of methods to assess their blood vessel function.
Period: Fresh Blood Transfusion
Arm/Group | Fresh Blood, Then Aged Blood
Started | 17
Completed | 17
Not Completed | 0
Period: Aged Blood Transfusion
Arm/Group | Fresh Blood, Then Aged Blood
Started | 17
Completed | 8
Not Completed | 9
Not completed — Withdrawal by Subject | 9

BASELINE CHARACTERISTICS:
Population: Only the 8 volunteers who completed both arms of this study are analyzed here.
Groups:
- All Subjects: Subjects donated one unit of blood, which was processed, stored for 3-5 days, then infused back to the subject (Fresh Blood). At least 8 weeks later, they returned, donated another unit of blood, which was stored for 40-42 days, then infused back to the subject (Aged Blood). Before and after each transfusion, the subjects was tested with a variety of methods to assess their blood vessel function.
Arm/Group | All Subjects
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.6 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Race/Ethnicity, Customized [Number; unit: participants] — The volunteer population was composed of 4 Caucasians, 1 African-American, 2 Asian-Americans, and 1 participant whose race was categorized as "other".
  participants
    Caucasian | 4
    African-American | 1
    Asian-American | 2
    "Other" | 1
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: The Effects of Storage-related RBC Changes on Acetylcholine-stimulated (NO-mediated) Forearm Blood Flow.
Description: The primary outcome measures are changes in forearm blood flow (FBF) in recipients of fresh or stored RBC transfusions in response to acetylcholine. Secondary measures include changes in FBF with acetylcholine with or without L-NMMA, and changes in FBF with forearm exercise. In addition, flow mediated dilation (FMD) measurements will also be used to assess changes in brachial artery diameter before and after fresh vs aged RBC transfusions.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: mL / 100 mL / min
Arm/Group | Fresh Blood, Then Aged Blood
Number analyzed (Participants) | 8
mL / 100 mL / min
  Prior to transfusion; fresh blood | 19.02 (8.22)
  Prior to transfusion; aged blood | 18.42 (4.73)
  Immediately after transfusion; fresh blood | 17.61 (4.8)
  Immediately after transfusion; aged blood | 22.89 (5.52)
  24 hours after transfusion; fresh blood | 22.83 (19.66)
  24 hours after transfusion; aged blood | 19.66 (3.62)

ADVERSE EVENTS:
Time Frame: Within 6 months of the start of the study.
Description: The occurrence of adverse events was based on observations of the study staff and/or volunteer self-reporting.
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

LIMITATIONS AND CAVEATS:
Primary limitation is that we are studying transfusion effects of fresh vs stored RBCs in healthy individuals, and not sick, anemic individuals as are often encountered in the hospital.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes